CLINICAL TRIAL: NCT07219290
Title: Pulmonary Function by Litter Position
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-45106
Record Dates: First submitted 2025-09-19; First posted 2025-10-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypothermia Due to Cold Environment; Trauma Patients
Keywords: search and rescue; pulmonary function; Suspension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flat (Active Comparator): Secured in a flat litter
  Interventions: Other: LItter position PFTs
- Vertical (Active Comparator): Secured in a vertical litter
  Interventions: Other: LItter position PFTs
- Pitched forward (Active Comparator): Secured in a litter leaning forward
  Interventions: Other: LItter position PFTs
- Baseline (Placebo Comparator): Sitting baseline pulmonary function
  Interventions: Other: LItter position PFTs

INTERVENTIONS:
Other: LItter position PFTs — Testing basic pulmonary function in three positions in a rescue litter, compared to sitting baseline

SUMMARY:
A litter is often needed to extract a person from an austere environment like the wilderness or from confined, urban spaces. A horizontal litter is generally assumed to be better for patient care, but often makes for a more difficult, if not impossible, evacuation from some settings such as confined space rescue, cave rescue, or wilderness rescue when the litter must be moved up or down a cliff with an undercut edge. A litter in a vertical orientation is easier to move in these situations, which may expedite movement towards definitive care. In some wilderness rescue circles, the mantra is that movement IS definitive care. It is already known that lying flat on the ground negatively affects pulmonary function compared to a sitting baseline.1 It is possible that a vertically oriented litter is better for a subset of patients with respiratory issues than a horizontal litter. The investigators hypothesize that pulmonary function measured by FEV1, FVC, and FEV1/FVC, is better in simulated patients in a vertically oriented litter compared to a horizontally oriented one.

DETAILED DESCRIPTION:
Objective To quantify changes in pulmonary function tests (PFTs) based on litter position.

Hypotheses:

* Compared to sitting baseline, all PFTs in the litter will have decreased forced vital capacity (FVC) and 1 second forced expiratory volume (FEV1).
* Compared to lying down, persons straight upright and pitched forward will have better forced vital capacity (FVC) and 1 second forced expiratory volume (FEV1).
* We do not hypothesize any changes in FEV1/FVC.

Study Design This randomized crossover study will use twelve healthy volunteers. All subjects will do baseline sitting pulmonary testing. Experimental order is balanced to avoid any training effects. Choice of sequence will be by random selection of envelope.

Methods Once consented, included subjects will do baseline sitting measurement of FEV1 and FVC which will give FEV1/FVC. Each subject will then be secured in a Ferno-Washington Model 71 litter wearing their own type 2 or 3 harness, or in a UL tested CMC ATOM Global Harness (California Mountain Corporation, Santa Barbara, CA) meeting ANSI Z359.11-2014 and NFPA 1983-2017 standards, if they don't have their own. The person will be secured with double Vs from the litter sides to the harness and footloops supporting them so their weight is on their feet and only minimally on the harness (if vertical). This process is consistent with industry standards for securing a patient in the litter and follows the specific model of the National Cave Rescue Commission.3 See figure 1 Prior to being secured in the litter the patient will do sitting baseline FEV1 and FVC with an NDDD spirograph. Once there is baseline data the subject will be secured in the litter. The investigators will then repeat spirometry, pulse, and blood pressure in a horizontal position (see figure 2), in a vertical position (see figure 3), and pitched slightly forward in a position that results from a Pike and Pivot rigging for raising up past a difficult cliff edge (see figure 4). The subject will get a rest period in their preferred position until pulse returns to within 5 beats of baseline.

Litter suspension will be with a four-legged litter spider when horizontal, with a high bridle tied directly to the litter head for the full vertical position, and from a low bridle in Pike-and-Pivot formation when pitched forward. The litter will be lifted into position with a 3:1 mechanical advantage system tied to an anchor. No matter the position, the lowest point of the litter will be no more than 6 inches off of the ground. The system will be configured for immediate lower for any expressed concern. The PI (RM) is a technical rescue instructor for the National Cave Rescue Commission and Assistant Training Officer-Technical Rescue for Fresno County search and rescue. The Co-PIs (SS and SD) are on the rope team of Fresno County search and rescue. Each is well versed in rope systems, anchor selection, and patient packaging.

ELIGIBILITY:
Inclusion Criteria:

* 130-310 pounds

Exclusion Criteria:

* Significant cardiac or pulmonary diseae

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity | Immediately
  Measurable lung volume on expiration

OTHER OUTCOMES:
FEV1 | Immediately
  Air volume exhaled in 1 second

CONTACTS AND LOCATIONS:
Overall Officials: Roger B Mortimer, MD, Principal Investigator — UCSF - Fresno
Locations (1):
- UCSF Fresno, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be submitted to a statistician
Supporting Information: Study Protocol, SAP
Time Frame: 1/1/26 to 6/1/26
Access Criteria: Roger Mortimer, MD Sarah Davis, DO Sue Spano, MD Amanda Mortimer, PhD